CLINICAL TRIAL: NCT03432416
Title: A Multicenter, Open-label Randomized Study on the Efficacy, Cycle Control and Safety of a Contraceptive Vaginal Ring Delivering a Daily Dose of Nestorone® and Estradiol (NES-E2 CVR).
Brief Title: Study of Efficacy, Cycle Control, and Safety of a NES-E2 Contraceptive Vaginal Ring
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCN012B
Record Dates: First submitted 2018-01-22; First posted 2018-02-14 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Women; Female Contraception
Keywords: Healthy Women; Female Contraception; Vaginal Ring; Contraceptive Vaginal Ring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen 1: Continuous Usage (Experimental): Contraceptive vaginal ring delivering a daily dose of Nestorone® and estradiol (NES-E2 CVR) worn continuously for 91 days.
  Interventions: Drug: NES-E2 CVR
- Regimen 2: Cyclical Usage (Experimental): Contraceptive vaginal ring delivering a daily dose of Nestorone® and estradiol (NES-E2 CVR) worn for 91 days, but is removed for 2 days each month (days 29-30, 59-60, and 90-91).
  Interventions: Drug: NES-E2 CVR

INTERVENTIONS:
Drug: NES-E2 CVR — NES-E2 CVR

SUMMARY:
This will be a multi-site, open-label, randomized clinical trial. The investigators will randomize 300 eligible participants in a 1:1 ratio to two different treatment regimens that are to be followed when using a contraceptive vaginal ring delivering a daily dose of Nestorone® and estradiol (NES-E2 CVR).

DETAILED DESCRIPTION:
The total duration of the study for each participant is expected to be approximately 13.5-15.5 months: including screening and enrollment (up to 8 weeks), 12 months of participation, and a post-removal follow up period removal of at least 17 days. After enrollment, subject visits occur at day 31, 92, 183, 274, and 364 with telephone calls at day 60, 120, 150, 210, 240, 300, and 330. Subjects will use a home pregnancy test 17 days post-removal of the ring and will call the site report the result and for safety follow-up. Another phone call will be required after that if the subject chooses not to being a hormonal contraceptive; this call will occur at the time of the subject's first spontaneous menses.

Subject recruitment is expected to begin Q1 (in the first quarter of) 2018 and is planned to continue through Q1 2019. However, if the enrollment rate declines, the enrollment period may be extended beyond this date. If this enrollment timeline is met, all subjects should finish active treatment by approximately the end of Q1 2020. The end of the study will occur when the last subject to be enrolled has completed her post-removal telephone call(s).

Preliminary results of the study are expected to be available Q3 of 2020 based on the current study plan.

ELIGIBILITY:
Inclusion Criteria:

1. Good general overall health with no chronic medical conditions that result in periodic exacerbations requiring significant medical care.
2. Age 18-35 years, inclusive, at the enrollment visit. (Note: subjects must be at least 18 years of age to provide consent.)
3. Have a regular menstrual cycle 21-35 days in duration when not using hormonal contraception
4. Have an intact uterus and at least one ovary.
5. Consistent use of effective contraception during the preceding cycle with no unprotected intercourse since last use (NOTE: women who use oral, transdermal, vaginal, or implantable hormonal contraceptives in the preceding cycle must have discontinued hormone use at least 4 days prior to start of treatment and must not have had unprotected intercourse since discontinuing the method. Copper IUD or Levonorgestrel releasing IUD users must have discontinued IUD use at least 4 days prior to start of treatment and have experienced a spontaneous menses following IUD removal.)
6. No use of injectable contraceptives (e.g. depomedroxyprogesterone acetate) during the 10 months prior to screening unless the subject has returned to normal menses (two consecutive menses) since last injection.
7. Have a negative pregnancy test at the enrollment visit.
8. Have a diastolic blood pressure (BP) <90 mm Hg and systolic BP <140 mm Hg after 5 minutes rest in sitting position at the admission visit (below hypertension stage 2). (Note: History of hypertension stage 2 or higher, even if controlled with treatment, is exclusionary.)
9. Willing to abstain from use of non-water based (including silicone based) vaginal lubricants during the study that could adversely affect the ring, causing it to expand.
10. Understand and sign an IRB-approved informed consent form prior to screening activities (including fasting blood draws).
11. BMI ≤ 35 kg/m2 and not having previously undergone bariatric surgery.
12. Planning to have at least one act of heterosexual intercourse without the use of another contraceptive method each month during study participation until end of treatment and at risk for pregnancy.

Exclusion Criteria:

1. Planning pregnancy during study participation through the end of treatment visit.
2. Within 30 days post-partum, currently breast-feeding, or has not had a spontaneous menses.
3. Post-abortal and has not had a spontaneous menses.
4. Abnormal genital bleeding.
5. Participating in another clinical trial involving an investigational product within the last 30 days (prior to screening) or planning to participate in another clinical trial during this study.
6. Not living in the catchment area of the study site.
7. Known hypersensitivity to progestins or estrogens.
8. Contraindications to combined estrogen-progestin contraceptive use including:

   1. Thrombophlebitis or thromboembolic disorders.
   2. Personal history of deep vein thrombophlebitis or thromboembolic disorders.
   3. History of venous thrombosis or embolism in a first-degree relative <55 years of age suggesting a familial defect in the blood coagulation system.
   4. History of thrombosis or embolism OR any other personal or family history which in the opinion of the investigator suggests increased risk.
   5. History of stroke.
   6. Known history of any of the following genetic mutations: Factor V Leiden mutation, prothrombin mutation, antithrombin deficiency, or other clinically significant thrombophilia.
   7. Known or suspected carcinoma of the breast.
   8. Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasm.
   9. History of cholestatic jaundice of pregnancy or jaundice with prior hormonal contraceptive use.
   10. History of hepatic adenomas or carcinomas.
   11. Known or suspected pregnancy.
   12. Smoking in women who are or will be 35 years during the course of the trial; women <35 years who smoke 15 cigarettes or more per day must be evaluated by the investigator for inclusion based on risk factors that would increase their risk for cardiovascular disease (CVD) and thromboembolism, e.g. lipid levels, glucose level, BP, BMI, family history of CVD at a young age. Individuals who use other forms of tobacco should be evaluated similarly by the investigator for inclusion based on the amount of tobacco use and their risk factors.
   13. History of retinal vascular lesions, unexplained partial or complete loss of vision.
   14. History of headaches with focal neurological symptoms (e.g., migraines with auras).
   15. Impaired mobility (e.g. wheelchair bound, bed-ridden) that, in the opinion of the investigator, places the woman at increased risk of thrombosis.
9. Unevaluated vaginal discharge or vaginal lesions. Subjects diagnosed at screening with a chlamydia or gonococcal infection may be included in the trial following treatment completion; partner treatment is also recommended. Subjects with yeast, trichomoniasis, or bacterial vaginosis infection requiring treatment may be enrolled after treatment completion. Investigators should determine if subjects are at an elevated risk for reinfection, e.g. multiple sex partners, untreated partner, and whether such subjects can be included. Women with a history of genital herpes can be included if outbreaks are infrequent.
10. Have a known clinically significant Pap test abnormality, as managed by normal standard of care guidelines, that would require repeat evaluation or treatment during study participation based on the initial Pap findings.
11. Known benign or malignant liver tumors, renal disease or active liver disease.
12. Invasive cancer (past history of any carcinoma or sarcoma, except non-melanoma skin cancer).
13. Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive.
14. Known or suspected current alcohol dependence, chronic marijuana use, or any illicit drug use that may affect metabolism/transformation of study product and/or study treatment compliance. A chronic marijuana user is defined as someone who uses marijuana 4 or more times per week for study purposes.
15. Elevated fasting clinical chemistry values or complete blood count (CBC) values designated clinically significant by the investigator or medically qualified sub-investigator.
16. Uncontrolled thyroid disease.
17. Known impaired hypothalamic-pituitary-adrenal axis.
18. Known hypersensitivity to silicone rubber.
19. History of toxic shock syndrome.
20. Vaginal anatomic abnormality such as cystocele or rectocele that would preclude correct use of a vaginal ring.
21. Planning major surgery during study participation.
22. Severe current constipation.
23. Use of liver enzyme inducers or inhibitors on a regular basis.
24. Known HIV infection.
25. Use of any medications, including antibiotics that can significantly interfere with the metabolism of hormonal contraceptives.
26. Have an anticipated need for regular condom use, defined as use of at least one condom per month after enrollment.
27. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.
28. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 385 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate | 1 year

SECONDARY OUTCOMES:
Change in subjects' bleeding patterns for continuous vs cyclic use as compared to reported baseline bleeding patterns when the subjects were not on hormonal contraception using a bleeding questionnaire. | 1 year
Difference in bleeding patterns for continuous vs cyclic use using a bleeding diary. | 1 year
Incidence of adverse events, including serious adverse events | 1 year
Summary of number of bleeding and spotting days per 30- and 90- day intervals using a bleeding diary. | Every 30 and 90 days up to a total of 1 year
Summary of cyclic versus continuous use adverse events. | 1 year
Summary of acceptability questionnaires. | 1 year
Changes in complete blood count (CBC) labs from study entry (baseline) | 1 year
Changes in fasting sodium from study entry (baseline) | 1 year
Changes in fasting potassium from study entry (baseline) | 1 year
Changes in fasting chloride from study entry (baseline) | 1 year
Changes in fasting HCO3/CO2 from study entry (baseline) | 1 year
Changes in fasting glucose from study entry (baseline) | 1 year
Changes in fasting creatinine from study entry (baseline) | 1 year
Changes in fasting blood urea nitrogen (BUN) from study entry (baseline) | 1 year
Changes in fasting calcium from study entry (baseline) | 1 year
Changes in fasting Gamma-glutamyl transferase or Gamma-glutamyl transpeptidase (GGTP) from study entry (baseline) | 1 year
Changes in fasting protein from study entry (baseline) | 1 year
Changes in fasting albumin from study entry (baseline) | 1 year
Changes in fasting total bilirubin from study entry (baseline) | 1 year
Changes in fasting direct bilirubin from study entry (baseline) | 1 year
Changes in fasting alkaline phosphatase (ALPH) from study entry (baseline) | 1 year
Changes in fasting Alanine Aminotransferase (ALT) from study entry (baseline) | 1 year
Changes in fasting Aspartate Aminotransferase (AST) from study entry (baseline) | 1 year
Changes in total cholesterol from study entry (baseline) | 1 year
Changes in triglycerides from study entry (baseline) | 1 year
Changes in high-density lipoprotein (HDL) from study entry (baseline) | 1 year
Changes in low-density lipoprotein (LDL) from study entry (baseline) | 1 year

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Essential Access Health, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Bellevue Hospital Center, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health Science University, Portland, Oregon
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daulaire N, Leidl P, Mackin L et al., Promises to Keep: The Toll of Unintended Pregnancies on Women's Lives in the Developing World. Washington, DC: Global Health Council; 2002; 11.
- [Background] Speidel JJ, Harper CC, Shields WC. The potential of long-acting reversible contraception to decrease unintended pregnancy. Contraception. 2008 Sep;78(3):197-200. doi: 10.1016/j.contraception.2008.06.001. Epub 2008 Jul 9. No abstract available. PMID 18692608
- [Background] Finer LB, Henshaw SK. Disparities in rates of unintended pregnancy in the United States, 1994 and 2001. Perspect Sex Reprod Health. 2006 Jun;38(2):90-6. doi: 10.1363/psrh.38.090.06. PMID 16772190
- [Background] Sitruk-Ware R. New progestagens for contraceptive use. Hum Reprod Update. 2006 Mar-Apr;12(2):169-78. doi: 10.1093/humupd/dmi046. Epub 2005 Nov 16. PMID 16291771
- [Background] Sitruk-Ware R. Pharmacological profile of progestins. Maturitas. 2008 Sep-Oct;61(1-2):151-7. doi: 10.1016/j.maturitas.2008.11.011. PMID 19434887
- [Background] Heikinheimo O, Ranta S, Moo-Young A, Lahteenmaki P, Gordon K. Parenteral administration of progestin Nestorone to lactating cynomolgus monkeys: an ideal hormonal contraceptive at lactation? Hum Reprod. 1999 Aug;14(8):1993-7. doi: 10.1093/humrep/14.8.1993. PMID 10438416
- [Background] Heikinheimo O, Noe G, Haukkamaa M, Lahteenmaki P. The progestin ST 1435--rapid metabolism in man. Contraception. 1994 Sep;50(3):275-89. doi: 10.1016/0010-7824(94)90073-6. PMID 7805378
- [Background] Kumar N, Koide SS, Tsong Y, Sundaram K. Nestorone: a progestin with a unique pharmacological profile. Steroids. 2000 Oct-Nov;65(10-11):629-36. doi: 10.1016/s0039-128x(00)00119-7. PMID 11108869
- [Background] Kumar N, Fagart J, Liere P, Mitchell SJ, Knibb AR, Petit-Topin I, Rame M, El-Etr M, Schumacher M, Lambert JJ, Rafestin-Oblin ME, Sitruk-Ware R. Nestorone(R) as a Novel Progestin for Nonoral Contraception: Structure-Activity Relationships and Brain Metabolism Studies. Endocrinology. 2017 Jan 1;158(1):170-182. doi: 10.1210/en.2016-1426. PMID 27824503
- [Background] Haukkamaa M, Laurikka-Routti M, Heikinheimo O, Moo-Young A. Contraception with subdermal implants releasing the progestin ST-1435: a dose-finding study. Contraception. 1992 Jan;45(1):49-55. doi: 10.1016/0010-7824(92)90140-o. PMID 1591921
- [Background] Fraser IS, Weisberg E, Brache V, Alvarez F, Massai R, Mishell DR Jr, Apter D, Gale J, Tsong YY, Sivin I. Serum Nestorone and ethinyl estradiol levels, and ovulation inhibition in women using three different dosage combinations of a Nestorone progestogen-ethinyl estradiol contraceptive vaginal ring on a bleeding-signaled regimen. Contraception. 2005 Jul;72(1):40-5. doi: 10.1016/j.contraception.2004.12.015. PMID 15964291
- [Background] Sivin I, Mishell DR Jr, Alvarez F, Brache V, Elomaa K, Lahteenmaki P, Massai R, Miranda P, Croxatto H, Dean C, Small M, Nash H, Jackanicz TM. Contraceptive vaginal rings releasing Nestorone and ethinylestradiol: a 1-year dose-finding trial. Contraception. 2005 Feb;71(2):122-9. doi: 10.1016/j.contraception.2004.08.010. PMID 15707562
- [Background] Weisberg E, Brache V, Alvarez F, Massai R, Mishell DR Jr, Apter D, Gale J, Sivin I, Tsong YY, Fraser IS. Clinical performance and menstrual bleeding patterns with three dosage combinations of a Nestorone progestogen/ethinyl estradiol contraceptive vaginal ring used on a bleeding-signaled regimen. Contraception. 2005 Jul;72(1):46-52. doi: 10.1016/j.contraception.2004.12.014. PMID 15964292
- [Background] Rad M, Kluft C, Menard J, Burggraaf J, de Kam ML, Meijer P, Sivin I, Sitruk-Ware RL. Comparative effects of a contraceptive vaginal ring delivering a nonandrogenic progestin and continuous ethinyl estradiol and a combined oral contraceptive containing levonorgestrel on hemostasis variables. Am J Obstet Gynecol. 2006 Jul;195(1):72-7. doi: 10.1016/j.ajog.2005.12.007. Epub 2006 Mar 20. PMID 16545330
- [Background] Kluft C, Meijer P, LaGuardia KD, Fisher AC. Comparison of a transdermal contraceptive patch vs. oral contraceptives on hemostasis variables. Contraception. 2008 Feb;77(2):77-83. doi: 10.1016/j.contraception.2007.10.004. Epub 2008 Jan 11. PMID 18226669
- [Background] Mashchak CA, Lobo RA, Dozono-Takano R, Eggena P, Nakamura RM, Brenner PF, Mishell DR Jr. Comparison of pharmacodynamic properties of various estrogen formulations. Am J Obstet Gynecol. 1982 Nov 1;144(5):511-8. doi: 10.1016/0002-9378(82)90218-6. PMID 6291391
- [Background] Marty JP, James M, Hajo N, Wepierre J Percutaneous absorption of oestradiol and progesterone: Pharmacokinetic studies. In P Mauvais-Jarvis, CFH Vickers, J Wepierre (Eds), Percutaneous absorption of steroids. London: Academic Press Inc. (London) Ltd. 1980.
- [Background] Timmer CJ, Mulders TM. Pharmacokinetics of etonogestrel and ethinylestradiol released from a combined contraceptive vaginal ring. Clin Pharmacokinet. 2000 Sep;39(3):233-42. doi: 10.2165/00003088-200039030-00005. PMID 11020137
- [Background] Jensen JT, Burke AE, Barnhart KT, Tillotson C, Messerle-Forbes M, Peters D. Effects of switching from oral to transdermal or transvaginal contraception on markers of thrombosis. Contraception. 2008 Dec;78(6):451-8. doi: 10.1016/j.contraception.2008.07.004. Epub 2008 Aug 28. PMID 19014790
- [Background] Sitruk-Ware R, Plu-Bureau G, Menard J, Conard J, Kumar S, Thalabard JC, Tokay B, Bouchard P. Effects of oral and transvaginal ethinyl estradiol on hemostatic factors and hepatic proteins in a randomized, crossover study. J Clin Endocrinol Metab. 2007 Jun;92(6):2074-9. doi: 10.1210/jc.2007-0026. Epub 2007 Mar 20. PMID 17374706
- [Background] Brache V, Mishell DR, Lahteenmaki P, Alvarez F, Elomaa K, Jackanicz T, Faundes A. Ovarian function during use of vaginal rings delivering three different doses of Nestorone. Contraception. 2001 May;63(5):257-61. doi: 10.1016/s0010-7824(01)00199-8. PMID 11448466
- [Background] Odlind V, Lithell H, Selinus I, Vessby B. Unaltered lipoprotein and carbohydrate metabolism during treatment with contraceptive subdermal implants containing ST-1435. Ups J Med Sci. 1984;89(2):151-8. doi: 10.3109/03009738409178475. PMID 6380075
- [Background] Goebelsmann U, Mashchak CA, Mishell DR Jr. Comparison of hepatic impact of oral and vaginal administration of ethinyl estradiol. Am J Obstet Gynecol. 1985 Apr 1;151(7):868-77. doi: 10.1016/0002-9378(85)90664-7. PMID 3920910
- [Background] Protocol 330. Clinical Study Report on File. Population Council, New York, NY.
- [Background] Archer DF, Jensen JT, Johnson JV, Borisute H, Grubb GS, Constantine GD. Evaluation of a continuous regimen of levonorgestrel/ethinyl estradiol: phase 3 study results. Contraception. 2006 Dec;74(6):439-45. doi: 10.1016/j.contraception.2006.07.005. Epub 2006 Sep 18. PMID 17157099
- [Background] Scarabin PY, Oger E, Plu-Bureau G; EStrogen and THromboEmbolism Risk Study Group. Differential association of oral and transdermal oestrogen-replacement therapy with venous thromboembolism risk. Lancet. 2003 Aug 9;362(9382):428-32. doi: 10.1016/S0140-6736(03)14066-4. PMID 12927428
- [Background] Belsey EM, Machin D, d'Arcangues C. The analysis of vaginal bleeding patterns induced by fertility regulating methods. World Health Organization Special Programme of Research, Development and Research Training in Human Reproduction. Contraception. 1986 Sep;34(3):253-60. doi: 10.1016/0010-7824(86)90006-5. PMID 3539509
- [Background] Merkatz RB, Plagianos M, Hoskin E, Cooney M, Hewett PC, Mensch BS. Acceptability of the Nestorone(R)/ethinyl estradiol contraceptive vaginal ring: development of a model; implications for introduction. Contraception. 2014 Nov;90(5):514-21. doi: 10.1016/j.contraception.2014.05.015. Epub 2014 Jun 2. PMID 24993487
- [Background] Isidori AM, Pozza C, Esposito K, Giugliano D, Morano S, Vignozzi L, Corona G, Lenzi A, Jannini EA. Development and validation of a 6-item version of the female sexual function index (FSFI) as a diagnostic tool for female sexual dysfunction. J Sex Med. 2010 Mar;7(3):1139-46. doi: 10.1111/j.1743-6109.2009.01635.x. Epub 2009 Dec 1. PMID 19968774
- [Background] Borch KH, Braekkan SK, Mathiesen EB, Njolstad I, Wilsgaard T, Stormer J, Hansen JB. Anthropometric measures of obesity and risk of venous thromboembolism: the Tromso study. Arterioscler Thromb Vasc Biol. 2010 Jan;30(1):121-7. doi: 10.1161/ATVBAHA.109.188920. Epub 2009 Oct 15. PMID 19834110
- [Background] Pomp ER, le Cessie S, Rosendaal FR, Doggen CJ. Risk of venous thrombosis: obesity and its joint effect with oral contraceptive use and prothrombotic mutations. Br J Haematol. 2007 Oct;139(2):289-96. doi: 10.1111/j.1365-2141.2007.06780.x. PMID 17897305
- [Background] Simmons KB, Kumar N, Plagianos M, Roberts K, Hoskin E, Han L, Alami M, Creasy G, Variano B, Merkatz R. Effects of concurrent vaginal miconazole treatment on the absorption and exposure of Nestorone(R) (segesterone acetate) and ethinyl estradiol delivered from a contraceptive vaginal ring: a randomized, crossover drug-drug interaction study. Contraception. 2018 Mar;97(3):270-276. doi: 10.1016/j.contraception.2017.10.010. Epub 2017 Oct 31. PMID 29097225